CLINICAL TRIAL: NCT03551522
Title: A Phase 2, Double-Blind, Randomized, Placebo-Controlled Study Followed by an Open-Label Extension Period to Evaluate the Activity of Seladelpar in Subjects With Nonalcoholic Steatohepatitis (NASH)
Brief Title: A Study to Evaluate Seladelpar in Subjects With Nonalcoholic Steatohepatitis (NASH)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: unexpected histological findings
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CB8025-21730
Record Dates: First submitted 2018-05-09; First posted 2018-06-11 (Actual); Results first posted 2022-07-05 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-07

CONDITIONS: NASH - Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — seladelpar; (2-methyl-4-(5-methyl-2-(4-trifluoromethyl-phenyl)-2H-(1,2,3)triazol-4-ylmethylsulfanyl)phenoxy)acetic acid

STUDY DESIGN:
Intervention Model Description: Randomization: 1:2:2:2 (placebo: seladelpar 10 mg: 20 mg: 50 mg)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind Placebo Controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Seladelpar 10 mg (Experimental): Subjects enrolled will receive seladelpar 10 mg, 20 mg, 50 mg or placebo daily for 52 weeks.
  Interventions: Drug: Seladelpar
- Seladelpar 20 mg (Experimental): Subjects enrolled will receive seladelpar 10 mg, 20 mg, 50 mg or placebo daily for 52 weeks.
  Interventions: Drug: Seladelpar
- Seladelpar 50 mg (Experimental): Subjects enrolled will receive seladelpar 10 mg, 20 mg, 50 mg or placebo daily for 52 weeks.
  Interventions: Drug: Seladelpar
- Placebo (Placebo Comparator): Subjects enrolled will receive seladelpar 10 mg, 20 mg, 50 mg or placebo daily for 52 weeks.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Seladelpar — 10 mg, 20 mg, or 50 mg
  Other Names: MBX-8025
  Arms: Seladelpar 10 mg; Seladelpar 20 mg; Seladelpar 50 mg
Drug: Placebos — Matching placebo Capsule
  Arms: Placebo

SUMMARY:
A Phase 2, Double-Blind (DB), Randomized, Placebo-Controlled Study Followed by an Open-Label Extension Period to Evaluate the Activity of Seladelpar in Subjects with Nonalcoholic Steatohepatitis (NASH)

OLE phase was not analyzed due to the early termination of the study

DETAILED DESCRIPTION:
Primary Objectives

1. To evaluate the effect of seladelpar on hepatic fat fraction, as assessed by magnetic resonance imaging-proton density fat fraction (MRI-PDFF) at Week 12 in the DB phase
2. To evaluate the safety and tolerability of seladelpar in the DB and OLE phases

Secondary Objectives

1. To evaluate the effect of seladelpar on MRI- PDFF at Week 26 and Week 52 in the DB phase
2. To evaluate the effect of seladelpar on histological improvement of nonalcoholic fatty liver disease activity score (NAS) at Week 52 in the DB phase
3. To evaluate the effect of seladelpar on histological improvement of fibrosis at Week 52 in the DB phase
4. To evaluate the effect of seladelpar on metabolic biochemical markers and biochemical markers of inflammation in the DB and OLE phases

ELIGIBILITY:
DB Inclusion Criteria:

1. Must be able to provide written informed consent (signed and dated) and any authorizations required by local law
2. 18 to 75 years old (inclusive)
3. Histological evidence of definite NASH on a liver biopsy (obtained during the screening period or historical liver biopsy obtained no more than 90 days prior to the initial screening visit)
4. NAS of 4 points or greater with a score of at least 1 point in each component (steatosis, lobular inflammation, and ballooning)
5. Fibrosis stage 1, 2, or 3 on liver biopsy
6. MRI-PDFF ≥ 10%
7. Females of reproductive potential must use at least one barrier contraceptive and a second effective birth control method during the study and for at least 30 days after the last dose of study drug. Male subjects who are sexually active with female partners of reproductive potential must use barrier contraception and their female partners must use a second effective birth control method during the study and for at least 90 days after the last dose of study drug.

DB Exclusion Criteria:

1. Significant alcohol consumption, defined as more than 2 drink units per day (equivalent to 20 g) in women and 3 drink units per day (equivalent to 30 g) in men, or inability to reliably quantify alcohol intake
2. Treatment with drugs associated with nonalcoholic fatty liver disease (NAFLD) (amiodarone, methotrexate, oral glucocorticoids at doses greater than 5 mg/day, tamoxifen, estrogens at doses greater than those used for hormone replacement or contraception, anabolic steroids (such as testosterone and valproic acid) for more than 4 weeks within the last 2 months prior to the initial screening
3. Treatment with pioglitazone or high-dose vitamin E (>400 IU/day) within the last 2 months prior to the initial screening
4. Initiation of treatment with a glucagon-like peptide-1 (GLP-1) agonist or a dose change within the last 2 months prior to the initial screening
5. Prior or planned bariatric surgery (a prior reversed sleeve gastrectomy is permitted)
6. Poorly controlled type 2 diabetes mellitus as defined by hemoglobin A1c [HbA1c] 9.5% or higher or type 1 diabetes mellitus
7. Diabetic patients who are taking sodium/glucose cotransporter 2 (SGLT-2) inhibitors must be on a stable dose within 2 months prior to the initial screening and throughout the study
8. Significant weight loss within the last 6 months (e.g., > 10%)
9. Use of any weight-loss medication for 3 months prior to and during the study period
10. Body mass index (BMI) < 18.5 kg/m2
11. Hepatic decompensation defined as the presence of any of the following:

    * Serum albumin less than 3.5 g/dL
    * International normalized ratio (INR) greater than 1.4 (unless due to therapeutic anticoagulants)
    * Total bilirubin greater than 2 mg/dL with the exception of Gilbert syndrome
    * History of esophageal varices, ascites, or hepatic encephalopathy
12. Other chronic liver diseases

    * Active hepatitis B as defined by presence of hepatitis B surface antigen (HBsAg)
    * Active hepatitis C as defined by presence of hepatitis C virus antibody (HCV AB) plus a positive HCV RNA
    * History or evidence of current active autoimmune hepatitis
    * History or evidence of primary biliary cholangitis (PBC)
    * History or evidence of primary sclerosing cholangitis
    * History or evidence of Wilson's disease
    * History or evidence of alpha-1-antitrypsin deficiency
    * History or evidence of hemochromatosis
    * History or evidence of drug-induced liver disease, as defined exposure and history
    * Known bile duct obstruction
    * Suspected or proven liver cancer
13. ALT > 200 U/L
14. AST < 20 U/L
15. Creatine kinase (CK) > upper limit of normal (ULN)
16. Serum creatinine > ULN
17. Platelet < lower limit of normal (LLN)
18. Inability to obtain a liver biopsy
19. History of biliary diversion
20. Known history of human immunodeficiency virus (HIV) infection
21. History of malignancy diagnosed or treated within 2 years

    * Recent localized treatment of squamous or non-invasive basal cell skin cancers is permitted
    * Cervical carcinoma in-situ is allowed if appropriately treated prior to Screening
    * Participants under active evaluation for malignancy are not eligible
22. Active substance abuse, based on Investigator judgment, including inhaled or injected drugs, within 1 year prior to the initial screening
23. Females who are pregnant or breastfeeding
24. Patients unable to undergo MRI-PDFF due to:

    * Contraindication to MRI examination
    * Severe claustrophobia impacting ability to perform MRI during the study, despite mild sedation/treatment with an anxiolytic
    * Weight or girth exceeds the scanner capacities
25. Treatment with any other investigational therapy or device within 30 days or within five half-lives, whichever is longer, prior to the initial screening
26. Active, serious medical disease with likely life expectancy < 5 years
27. Any other condition(s) that would compromise the safety of the subject or compromise study quality as judged by the Investigator

OLE Phase Enrollment Criteria

Subjects must fulfill the following before allowing to start OLE dosing:

1. Provide informed consent on or before Day 1 and prior to any OLE-related study procedures.
2. Completed through the Week 52 biopsy and Week 56 lab assessments in the DB phase
3. Meet the above DB phase Inclusion and Exclusion Criteria before Day 1 of the OLE phase, with the exception of the following:

   * AST < 20 U/L
   * Inability to obtain a liver biopsy (no new biopsy required for OLE)
   * Unable to undergo MRI-PDFF (no imaging performed in OLE)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2019-05-08 (Actual); Study Completion 2020-08-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - CymaBay Research Site, Glendale, Arizona
  - CymaBay Research Site, Tucson, Arizona
  - CymaBay Research Site, Los Angeles, California
  - CymaBay Research Site, Boca Raton, Florida
  - CymaBay Research Site, Lakewood Rch, Florida
  - CymaBay Research Site, Flowood, Mississippi
  - CymaBay Research Site, Clarksville, Tennessee
  - CymaBay Research Site, Germantown, Tennessee
  - CymaBay Research Site, Hermitage, Tennessee
  - CymaBay Research Site, Knoxville, Tennessee
  - CymaBay Research Site, Chandler, Texas
  - CymaBay Research Site, Dallas, Texas
  - CymaBay Research Site, Live Oak, Texas
  - CymaBay Research Site, Rollingwood, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alkhouri N, Beyer C, Shumbayawonda E, Andersson A, Yale K, Rolph T, Chung RT, Vuppalanchi R, Cusi K, Loomba R, Pansini M, Dennis A. Decreases in cT1 and liver fat content reflect treatment-induced histological improvements in MASH. J Hepatol. 2025 Mar;82(3):438-445. doi: 10.1016/j.jhep.2024.08.031. Epub 2024 Sep 25. PMID 39326675
- [Derived] Beyer C, Hutton C, Andersson A, Imajo K, Nakajima A, Kiker D, Banerjee R, Dennis A. Comparison between magnetic resonance and ultrasound-derived indicators of hepatic steatosis in a pooled NAFLD cohort. PLoS One. 2021 Apr 1;16(4):e0249491. doi: 10.1371/journal.pone.0249491. eCollection 2021. PMID 33793651

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: DB Phase: A total of 181 subjects were randomly assigned to receive placebo, seladelpar 10 mg/day, seladelpar 20 mg/day, or seladelpar 50 mg/day (1:2:2:2 ratio). Subjects were stratified by diabetic status (yes/no) and fibrosis stage (F1 versus F2-3). Study drug (placebo or seladelpar) was taken in a blinded manner orally once a day for a period of 52 weeks.
  OLE Phase: All subjects will receive seladelpar 50 mg regardless of dose received during the DB phase.
Groups:
- Period 1: Seladelpar 10 mg: DB Phase. Subjects were randomized to receive seladelpar 10 mg daily for 52 weeks.
- Period 1: Seladelpar 20 mg: DB Phase. Subjects were randomized to receive seladelpar 20 mg daily for 52 weeks.
- Period 1: Seladelpar 50 mg: DB Phase. Subjects were randomized to receive seladelpar 50 mg daily for 52 weeks.
- Period 1: Placebo: DB Phase. Subjects were randomized to receive placebo daily for 52 weeks.
- Period 2: Seladelpar 50 mg: OLE phase: All subjects received seladelpar 50 mg
Period: DB Phase
Arm/Group | Period 1: Seladelpar 10 mg | Period 1: Seladelpar 20 mg | Period 1: Seladelpar 50 mg | Period 1: Placebo | Period 2: Seladelpar 50 mg
Started | 53 | 51 | 50 | 27 | 0
Completed | 27 | 34 | 32 | 17 | 0
Not Completed | 26 | 17 | 18 | 10 | 0
Period: OLE Phase
Arm/Group | Period 1: Seladelpar 10 mg | Period 1: Seladelpar 20 mg | Period 1: Seladelpar 50 mg | Period 1: Placebo | Period 2: Seladelpar 50 mg
Started | 0 | 0 | 0 | 0 | 12
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 12

BASELINE CHARACTERISTICS:
Groups:
- Seladelpar 10 mg; Seladelpar 20 mg; Seladelpar 50 mg: Subjects were randomized to receive seladelpar 10 mg, 20 mg, 50 mg or placebo daily for 52 weeks.
  Seladelpar: 10 mg, 20 mg, or 50 mg
- Placebo: Subjects were randomized to receive seladelpar 10 mg, 20 mg, 50 mg or placebo daily for 52 weeks.
  Placebos: Matching placebo Capsule
- Total: Total of all reporting groups
Arm/Group | Seladelpar 10 mg | Seladelpar 20 mg | Seladelpar 50 mg | Placebo | Total
Number analyzed (Participants) | 53 | 51 | 50 | 27 | 181
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (12.48) | 56.6 (11.74) | 53.7 (11.18) | 53.9 (10.27) | 54.4 (11.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 35 | 33 | 18 | 122
  Male | 17 | 16 | 17 | 9 | 59
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 50 | 47 | 49 | 27 | 173
  Black or African American | 1 | 1 | 0 | 0 | 2
  Asian | 1 | 1 | 1 | 0 | 3
  American Indian or Alaska native | 1 | 1 | 0 | 0 | 2
  Multiple | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 53 | 51 | 50 | 27 | 181

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in Magnetic Resonance Imaging-proton Density Fat Fraction (MRI-PDFF)
Description: Evaluate the effect of seladelpar on hepatic fat fraction, as assessed by magnetic resonance imaging-proton density fat fraction (MRI-PDFF) at Week 12 in the double-blind (DB) phase.
  MRI-PDFF Relative (Percent) Change From Baseline to Week 12 - ANCOVA - mITT Population MRI-PDFF exam was used to quantify the hepatic proton density fat fraction noninvasively. The fat fraction is the proportion of mobile protons in liver tissue attributable to fat and thus, is a noninvasive magnetic resonance-based biomarker of liver triglyceride concentration.
Time Frame: Week 12
Population: mITT Population: defined as any subject who was randomized, received at least one dose of study drug, and had Baseline and Week 12 MRI-PDFF.
Measure: Least Squares Mean (Standard Error); unit: percentage of change from Baseline
Arm/Group | Seladelpar 10 mg | Seladelpar 20 mg | Seladelpar 50 mg | Placebo
Number analyzed (Participants) | 50 | 47 | 48 | 26
percentage of change from Baseline | -9.76 (4.153) | -14.24 (4.329) | -13.00 (4.305) | -20.78 (5.555)
Statistical Analysis 1: Comparison: Seladelpar 10 mg vs Placebo; Test type: Other — The LS Means, confidence intervals, and p-values come from an ANCOVA model with relative (percent) change from baseline as the dependent variable and treatment and stratification groups (diabetic status and fibrosis stage) as factors and baseline as a covariate; p = 0.0874, ANCOVA; LS Mean of Difference = 11.02, 95% CI 2-sided [-1.63 to 23.67]
Statistical Analysis 2: Comparison: Seladelpar 20 mg vs Placebo; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.3151, ANCOVA; LS Mean of Difference = 6.54, 95% CI 2-sided [-6.28 to 19.37]
Statistical Analysis 3: Comparison: Seladelpar 50 mg vs Placebo; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.2313, ANCOVA; LS Mean of Difference = 7.78, 95% CI 2-sided [-5.01 to 20.58]

2. Secondary Outcome: Percentage of Participants With Improvement of 2 Points or More in the Nonalcoholic Fatty Liver Disease Activity Score (NAS)
Description: Histopathology nonalcoholic fatty liver disease activity score (NAS) change from baseline ≤-2 (Improvements of 2 points or more in NAS) - mITT Population Total NAS score represents the sum of scores for steatosis, lobular inflammation, and ballooning, and ranges from 0-8. Diagnosis of NASH (or, alternatively, fatty liver not diagnostic of NASH) should be made first, then NAS is used to grade activity. NAS scores of 0-2 occurred in cases largely considered not diagnostic of NASH, scores of 3-4 were evenly divided among those considered not diagnostic, borderline, or positive for NASH. Scores of 5-8 occurred in cases that were largely considered diagnostic of NASH
Time Frame: Week 52
Population: mITTb population: The mITTb population is defined as any subject who is randomized, receives at least one dose of study drug, and has Baseline and Week 52/ET liver biopsies.
Measure: Number; unit: Percentage of Participants
Arm/Group | Seladelpar 10 mg | Seladelpar 20 mg | Seladelpar 50 mg | Placebo
Number analyzed (Participants) | 39 | 42 | 46 | 25
Percentage of Participants | 23.1 | 45.2 | 37.0 | 32.0

3. Secondary Outcome: Percent Change From Baseline in Alanine Aminotransferase (ALT) at Week 12 and Week 52
Description: Alanine Aminotransferase (ALT) Relative (percent) change of from Baseline to Weeks 12 and Week 52 - mITT Population A decreased serum levels of alanine aminotransferase (ALT) is a marker of liver function improvement.
Time Frame: Week 12, Week 52
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage of change from Baseline
Arm/Group | Seladelpar 10 mg | Seladelpar 20 mg | Seladelpar 50 mg | Placebo
Number analyzed (Participants) | 39 | 42 | 46 | 25
percentage of change from Baseline
  Week 12 | -24.05 (4.154) | -32.92 (4.075) | -38.29 (3.907) | -9.57 (5.034)
  Week 52 | -28.60 (5.044) | -43.93 (4.844) | -40.60 (4.682) | -2.26 (6.252)

4. Secondary Outcome: Percent Change From Baseline in Aspartate Aminotransferase (AST) at Week 12 and Week 52
Description: Relative (Percent) Change of Aspartate Aminotransferase (AST) From Baseline to Weeks 12 and Week 52 - mITT Population A decreased serum levels of Aspartate Aminotransferase (AST) is a marker of liver function improvement.
Time Frame: Weeks 12, Week 52
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage of change from baseline
Arm/Group | Seladelpar 10 mg | Seladelpar 20 mg | Seladelpar 50 mg | Placebo
Number analyzed (Participants) | 39 | 42 | 46 | 25
percentage of change from baseline
  Week 12 | -14.02 (4.793) | -16.03 (4.686) | -17.88 (4.491) | -14.75 (5.834)
  Week 52 | -20.62 (5.988) | -26.43 (5.698) | -18.43 (5.536) | -4.54 (7.490)

5. Secondary Outcome: Percent Change From Baseline in Gamma Glutamyl Transferase (GGT) at Week 12 and Week 52
Description: Relative (Percent) Change of Gamma Glutamyl Transferase (GGT) From Baseline to Weeks 12 and Week 52 - mITT Population A decreased serum levels of Gamma Glutamyl Transferase (GGT) is a marker of liver function improvement.
Time Frame: Weeks 12, Week 52
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percentage of change from Baseline
Arm/Group | Seladelpar 10 mg | Seladelpar 20 mg | Seladelpar 50 mg | Placebo
Number analyzed (Participants) | 39 | 42 | 46 | 25
Percentage of change from Baseline
  Week 12 | -28.67 (3.848) | -37.78 (3.760) | -42.50 (3.626) | -6.40 (4.630)
  Week 52 | -27.93 (5.674) | -45.84 (5.401) | -35.11 (5.255) | 0.71 (7.093)

6. Secondary Outcome: Number of Participants With Decrease in MRI-PDFF ≥ 30% From Baseline at Week 12 and Week 52
Description: Number of Participants with a relative decrease in MRI-PDFF ≥30% (ie, percent change ≥ 30%) at Weeks 12, and 52/ET (Early Termination) in the DB phase - mITT Population.
  MRI-PDFF exam was used to quantify the hepatic proton density fat fraction noninvasively. The fat fraction is the proportion of mobile protons in liver tissue attributable to fat and thus, is a noninvasive magnetic resonance-based biomarker of liver triglyceride concentration.
  MRI-PDFF response defined as ≥30% relative decline in MRI-PDFF is associated with ≥1 stage improvement in fibrosis and may be used as a surrogate marker of fibrosis regression in early phase clinical trials for NASH
Time Frame: Week 12, Week 52
Population: mITT Population: defined as any subject who is randomized, receives at least one dose of study drug, and has Baseline and Week 12 MRI-PDFF
Measure: Count of Participants; unit: Participants
Arm/Group | Seladelpar 10 mg | Seladelpar 20 mg | Seladelpar 50 mg | Placebo
Number analyzed (Participants) | 50 | 47 | 48 | 26
Participants
  Week 12 | 12 | 12 | 9 | 8
  Week 52/ET | 8 | 19 | 8 | 5

7. Secondary Outcome: Percentage Change From Baseline in Magnetic Resonance Imaging-proton Density Fat Fraction (MRI-PDFF) at Week 52
Description: Percentage Change from Baseline in MRI-PDFF to Weeks 52//ET - mITT Population MRI-PDFF exam was used to quantify the hepatic proton density fat fraction noninvasively. The fat fraction is the proportion of mobile protons in liver tissue attributable to fat and thus, is a noninvasive magnetic resonance-based biomarker of liver triglyceride concentration.
Time Frame: Week 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percentage of change from Baseline
Arm/Group | Seladelpar 10 mg | Seladelpar 20 mg | Seladelpar 50 mg | Placebo
Number analyzed (Participants) | 50 | 47 | 48 | 26
percentage of change from Baseline | -9.76 (27.323) | -23.98 (30.666) | -7.99 (30.650) | -18.30 (27.872)

8. Secondary Outcome: Number of Liver Biopsy Responders With Reversal of NASH Reversal of NASH (Ballooning Score of 0 and Lobular Inflammation Score of 0 or 1) and no Worsening of Hepatic Fibrosis at Week 52
Description: Liver Biopsy Responders with reversal of NASH (ballooning score of 0 and lobular inflammation score of 0 or 1 and no worsening of hepatic fibrosis) at Week 52/ET.
  The reversal of NASH was defined as the absence of hepatocellular ballooning (score of 0) and no or minimal inflammation (lobular inflammation score of 0 or 1).
Time Frame: Week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Seladelpar 10 mg | Seladelpar 20 mg | Seladelpar 50 mg | Placebo
Number analyzed (Participants) | 39 | 42 | 46 | 25
Participants | 4 | 8 | 12 | 2

9. Secondary Outcome: Percentage of Participants With Improvement by at Least 1 Stage in Fibrosis From Baseline at Week 12 and Week 52
Description: Proportion of subjects with improvement by at least 1 stage in fibrosis without worsening of NASH (ie, improvement by at least 1 fibrosis stage without worsening of NAS) at Week 52/ET - Cochran-Mantel-Haenszel - mITTb Population There five liver fibrosis stages (F0: no scarring (no fibrosis); F1: minimal scarring; F2: scarring has occurred and extends outside the liver area (significant fibrosis); F3: fibrosis spreading and forming bridges with other fibrotic liver areas (severe fibrosis); F4: cirrhosis or advanced scarring)
Time Frame: Week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Seladelpar 10 mg | Seladelpar 20 mg | Seladelpar 50 mg | Placebo
Number analyzed (Participants) | 39 | 42 | 46 | 25
Participants | 9 | 10 | 17 | 5

ADVERSE EVENTS:
Time Frame: Through DB Phase (from first dose of DB phase study drug, and up to 30 days after last dose of DB phase study drug or 1 day before the first dose of OLE phase, whichever was earlier), up to 56 weeks. AEs are only summarized in DB phase, not OLE phase.
Groups:
- Seladelpar 10 mg: Subjects were randomized to receive seladelpar 10 mg daily for 52 weeks.
  AEs are only summarized in DB phase, not OLE phase.
- Seladelpar 20 mg: Subjects were randomized to receive seladelpar 20 mg daily for 52 weeks.
  AEs are only summarized in DB phase, not OLE phase.
- Seladelpar 50 mg: Subjects were randomized to receive seladelpar 50 mg daily for 52 weeks.
  AEs are only summarized in DB phase, not OLE phase.
- Placebo: Subjects were randomized to receive placebo daily for 52 weeks.
  AEs are only summarized in DB phase, not OLE phase.
Arm/Group | Seladelpar 10 mg | Seladelpar 20 mg | Seladelpar 50 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/51 | 0/50 | 0/27
Serious Adverse Events (participants affected / at risk) | 1/53 | 3/51 | 5/50 | 0/27
Other Adverse Events (participants affected / at risk) | 45/53 | 49/51 | 48/50 | 25/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Seladelpar 10 mg (N=53) | Seladelpar 20 mg (N=51) | Seladelpar 50 mg (N=50) | Placebo (N=27)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gastroenteritis Escherichia coli (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Seladelpar 10 mg (N=53) | Seladelpar 20 mg (N=51) | Seladelpar 50 mg (N=50) | Placebo (N=27)
Cataract (Eye disorders) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (3) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 4 (4) | 3 (3) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 6 (7) | 4 (4) | 3 (3) | 3 (3)
Constipation (Gastrointestinal disorders) | 3 (3) | 4 (4) | 5 (5) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 6 (6) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (4) | 4 (4) | 3 (3) | 3 (3)
Nausea (Gastrointestinal disorders) | 7 (9) | 8 (9) | 6 (7) | 4 (4)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 4 (4) | 3 (3) | 2 (3)
Fatigue (General disorders) | 4 (4) | 3 (3) | 3 (3) | 2 (3)
Bronchitis (Infections and infestations) | 1 (1) | 4 (4) | 1 (1) | 1 (2)
Influenza (Infections and infestations) | 2 (2) | 3 (3) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 4 (5) | 1 (1)
Sinusitis (Infections and infestations) | 3 (3) | 2 (2) | 2 (2) | 2 (3)
Tooth infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 5 (8) | 2 (2) | 4 (5) | 3 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 5 (8) | 6 (8) | 3 (4)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 5 (6) | 3 (3) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 8 (10) | 2 (2) | 6 (6) | 4 (5)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 7 (7) | 4 (5) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (6) | 2 (2) | 4 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 3 (5) | 5 (5) | 2 (2) | 2 (3)
Headache (Nervous system disorders) | 6 (6) | 10 (10) | 2 (2) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1) | 2 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (4) | 3 (3) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) | 4 (4) | 0 (0)
Hypertension (Vascular disorders) | 6 (6) | 2 (2) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-12-20): https://cdn.clinicaltrials.gov/large-docs/22/NCT03551522/Prot_002.pdf
  • Statistical Analysis Plan (2020-02-28): https://cdn.clinicaltrials.gov/large-docs/22/NCT03551522/SAP_001.pdf